CLINICAL TRIAL: NCT03565302
Title: Gender-specific Role of the beta2-adrenergic Stimulation With Short- or Long-acting Selective Agonist in Relation to Muscle Remodelling, Function, Performance, and Anti-doping
Brief Title: Beta2-adrenergic Agonism and Muscle Remodelling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: FOR/TER
Record Dates: First submitted 2018-06-07; First posted 2018-06-21 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Hypertrophy; Physiologic Hypertrophy; Physical Activity
Keywords: Proteome; VO2max; Muscle function; Exercise performance; Skeletal muscle; Doping; Anti-Doping; Enantiomeric analysis
MeSH Terms: conditions — Hypertrophy; Motor Activity | interventions — Formoterol Fumarate; Terbutaline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): Subjects receive placebo treatment
  Interventions: Other: Placebo
- Long acting beta2-agonist (Experimental): Subjects are treated with long-acting beta2-agonist formoterol
  Interventions: Drug: Formoterol
- Short acting beta2-agonist (Experimental): Subjects are treated with short-acting beta2-agonist terbutaline
  Interventions: Drug: Terbutaline

INTERVENTIONS:
Drug: Formoterol — Subjects are treated with daily inhalation of formoterol
  Arms: Long acting beta2-agonist
Drug: Terbutaline — Subjects are treated with daily inhalation of terbutaline
  Arms: Short acting beta2-agonist
Other: Placebo — Subjects are treated with placebo
  Arms: Control

SUMMARY:
The study aims to investigate gender-specific adaptations to beta2-adrenoceptor stimulation with selective short- and long-acting beta2-agonist with emphasis on skeletal muscle in relation to performance enhancing effects and anti-doping

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, aged 18-45 years
* VO2max >55 ml/kg/min for men and >50 ml/kg/min for women (± biologic and techinical variation of 5.6% (Katch et al. 1982)
* Body Mass Index (BMI) < 26

Exclusion Criteria:

* Chronic user of beta2-agonist or allergy towards study drugs
* Serious adverse side effects of the used study drug
* Chronic disease that by the project physician would affect any of the outcomes of the study
* Smoker
* Chronic use of prescription medication (other than contraceptives for women)
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Proteome enrichment | Baseline and 6 weeks
  Change in enrichment (measured in muscle biopsies and assessed using GO annotations)

SECONDARY OUTCOMES:
Body composition | Baseline, 2 weeks, 4 weeks and 6 weeks
  Change in body composition (measured by dual energy x ray absorptiometry)
Maximal oxygen consumption (VO2max) | Baseline, 2 weeks, 4 weeks and 6 weeks
  Change in VO2max (measured during bike ergometer cycling to exhaustion)

OTHER OUTCOMES:
Drug exposure | Day 1-14 and day 49-56
  Measured in urine using enantiomeric analysis

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided